CLINICAL TRIAL: NCT07088588
Title: A First-in-Human Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of SYN608, a Poly ADP-ribose Glycohydrolase (PARG) Inhibitor in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of SYN608 for the Treatment of Advanced or Metastatic Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou SynRx Therapeutics Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYN-608-101
Record Dates: First submitted 2025-07-18; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Cancer; Metastatic Solid Tumor; Ovarian Cancer; Breast Cancer; BRCA Mutation; HRR Deficiency
MeSH Terms: conditions — Neoplasm Metastasis; Ovarian Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SYN608 tablet (Experimental): SYN608 tablet monotherapy
  Interventions: Drug: SYN608

INTERVENTIONS:
Drug: SYN608 — Patients will orally receive SYN608

SUMMARY:
This interventional study will evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary efficacy of SYN608 as monotherapy in adult patients with advanced solid tumors

DETAILED DESCRIPTION:
This study is a Phase I, open-label, multicentre study of SYN608 administered orally in patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Having signed the written Informed Consent Form (ICF);
* Male or female aged ≥18 years;
* Life expectancy ≥12 weeks;
* Eastern Cooperative Oncology Group (ECOG) Performance Score 0 or 1;
* Patients with histologically or cytologically confirmed locally advanced or metastatic breast cancer, ovarian cancer or other advanced solid tumors who have experienced disease progression, and available standard of care (SOC) therapies had been exhausted;
* be willing to provide tumor tissue samples (fresh frozen [SF] or previously retained paraffin-embedded [FFPE] tumor tissue samples) or peripheral blood germline DNA or ctDNA sample to detect BRCA mutation, or other deficiency in the Homologous Recombination (HR) pathway (by the detection method of next generation sequencing [NGS])
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1;
* No serious hematological, cardiopulmonary, or liver or kidney diseases other than the primary disease;
* Adequate organ function and bone marrow function.

Exclusion Criteria:

* Previous or current use of Poly (ADP) ribose glycohydrolase (PARG) inhibitors;
* Serious allergy to the study drug or any of its excipients;
* Current or previous other malignancy unless treated radically and with no evidence of recurrence or metastasis within the past 5 years;
* Central nervous system (CNS) metastasis or meningeal metastasis with clinical symptoms, or other evidence indicating that CNS metastasis or meningeal metastasis has not been adequately controlled;
* Patients with Myelodysplastic syndrome (MDS)/Acute myeloid leukemia (AML) or with features suggestive of MDS/AML;
* Dysphagia or refractory nausea and vomiting, malabsorption, extracorporeal biliary shunts, or gastrointestinal disorders that affect drug absorption, e.g., Crohn's disease, ulcerative colitis, or short bowel syndrome, or other malabsorption conditions;
* Treatment with an anti-cancer small molecule within 5 half-lives (t1/2), or 2 weeks, whichever is shorter;
* History of use within 2 weeks prior to the first dose of the study treatment and need to use protocol-prohibited potent inhibitors or potent inducers of cytochrome P450 (CYP) 3A4/BCRP/P-gp during the study;
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease;
* Serious systemic diseases or laboratory abnormalities or other conditions that, at the Investigator's discretion, will make it unsuitable for the patient to participate in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 105 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 3 years
  MTD is defined as the maximum dose level at which ≤1 patient have dose limiting toxicities (DLTs) during the DLT observation period, and it should be determined with 6 evaluable patients.
Number of participants with Dose Limiting Toxicities (DLTs) | From first dose of study treatment until the end of Cycle 1 (each cycle is 21-days)
  Severity of adverse events as assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Number of participants experiencing adverse events (AEs)/serious adverse events (SAEs) | From time of information consent to 30 days post last dose, up to 3 years
  Number of participants with incidence of adverse events and with serious adverse events including changes from baseline in laboratory parameters, vital signs, Electrocardiogram (ECG), and physical examination, etc.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters | Up to 3 years
  To characterize the PK Peak Plasma Concentration (Cmax) of SYN608 monotherapy
Pharmacokinetic (PK) parameters | Up to 3 years
  To characterize the PK Time to Peak drug Concentration (Tmax) of SYN608 monotherapy
Pharmacokinetic (PK) parameters | Up to 3 years
  To characterize the PK Area under the plasma concentration versus time curve (AUC) of SYN608
Pharmacokinetic (PK) parameters | Up to 3 years
  To characterize the PK profile of SYN608 by measuring elimination half-life (t1/2)
Objective Response Rate (ORR) | Up to 3 years
  ORR is defined as proportion of patients who achieved complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 recorded from first investigational product treatment until disease progression or death due to any cause. The confirmation of response for patients who has PR or CR at first time should be performed by at least 4 weeks. For castration-resistant prostate cancer (CRPC) patients, bone lesion will be assessed according to Prostate Cancer Working Group 3 (PCWG3) criteria.
Duration of Response (DoR) and Time to Response (TTR) | Up to 3 years
  DOR is defined, for patients with an objective response, as the time from first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression or death due to any cause.
Progression Free Survival (PFS) | Up to 3 years
  PFS is defined as the time from the first study treatment to the date of the first documentation of objective progression of disease (PD) or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - FuDan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai GoBroad Cancer Hospital China Pharmaceutical University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No